CLINICAL TRIAL: NCT03949998
Title: The Immediate Effects of Dry Needling on Post-concussion Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Dr. Margo Mountjoy, Adjunct Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-02-035
Record Dates: First submitted 2019-04-29; First posted 2019-05-14 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Post-Concussive Syndrome, Chronic
Keywords: Dry Needling
MeSH Terms: conditions — Post-Concussion Syndrome | interventions — Dry Needling; Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dry Needling (Experimental): Participants will receive dry needling of the following muscles as indicated: upper fibres trapezius, levator scapulae, cervical multifidus, suboccipitals.
  Interventions: Device: Dry Needling
- Dry Needling + Manual Therapy (Active Comparator): Participants will receive dry needling of the following muscles as indicated: upper fibres trapezius, levator scapulae, cervical multifidus, suboccipitals IN ADDITION TO manual therapy of the above muscles and/or cervical joint traction and/or mobilization as indicated.
  Interventions: Device: Dry Needling; Other: Manual Therapy
- Manual Therapy (Active Comparator): Participants will receive manual therapy of the following muscles as indicated: upper fibres trapezius, levator scapulae, cervical multifidus, suboccipitals and/or cervical joint traction and/or mobilization as indicated.
  Interventions: Other: Manual Therapy

INTERVENTIONS:
Device: Dry Needling — Comparison between dry needling and/or manual therapy of the cervical region.
  Other Names: Intramuscular Stimulation (Gunn IMS); Integrated Dry Needling (IDN)
  Arms: Dry Needling; Dry Needling + Manual Therapy
Other: Manual Therapy — soft tissue release, cervical traction and/or cervical mobilization
  Arms: Dry Needling + Manual Therapy; Manual Therapy

SUMMARY:
In about 15% of adult concussion cases, symptoms last longer than 2 weeks and can largely impact the individual's ability to work, be physically active and participate in everyday life. These symptoms are often partially related to unresolved neck muscle tightness and other neck-related symptoms. Dry needling is a technique that uses acupuncture needles to release muscle knots, decrease neck muscle tightness and decrease neck pain. As far as the investigators are aware, there have been no studies looking at the effects of dry needling on symptoms of chronic concussion. This study will compare the effects of dry needling to traditional hands-on physiotherapy treatment of the neck for concussion-related symptoms. Participants with chronic concussion symptoms will receive either dry needling, hands-on manual physiotherapy or both. Concussion symptoms, symptom severity, neck range of motion and pain with pressure over neck muscles will be compared before and after treatment, and the day after treatment. The investigators expect that the greatest improvement in all of these will be seen in the group receiving both interventions, both immediately after treatment and the following day. If dry needling can immediately improve concussion symptoms, patients may better tolerate therapeutic exercise and experience quicker resolution of chronic symptoms.

DETAILED DESCRIPTION:
All participants will be tested in clinic once, for approximately a half hour. For all groups, outcome measures relating to concussion symptoms, cervical range of motion and pain pressure thresholds will be taken prior to and after the intervention.

In the DN group, four muscles (upper fibres trapezius, cervical multifidus, levator scapulae and suboccipitals) will be palpated by a physiotherapist trained in dry needling. If a palpable trigger point is found, the physiotherapist will perform dry needling until a local twitch response is elicited. If a trigger point is not found, no dry needling will take place. In this way, up to 8 total muscles will be needled during the session. The participant will be in prone for the above procedure.

In the MT group, soft tissue release will be performed on the above four muscles bilaterally. Cervical traction (unilateral grade 3 oscillatory distraction technique, any cervical segment between C0/C1 and C7/C7, 3-5 sets of 30 seconds) and mobilization (unilateral inferior-medial-posterior or superior-anterior-lateral, grade 3 oscillatory, any cervical segment between C0/C1 and C7/C7, 3-5 sets of 30 seconds ) will also be performed if the physiotherapist deems it necessary, specific to the spinal level noted to be involved. In the DN+MT group, MT interventions will be performed first, followed by DN, of the four above muscles. Immediately following intervention, the outcome measures will all be re-tested. The participants will also be instructed to fill out the SCAT-5 Step 2 upon waking the next morning. Additionally, if one or more of the cervical motions caused pain during initial testing, they will be asked to repeat the motion and report the current level of pain on the VAS scale.

ELIGIBILITY:
Inclusion Criteria:

* experiencing concussion symptoms at least 4 weeks following an external impact injury to the head

Exclusion Criteria:

* medical diagnoses of depression and/or anxiety
* skull fractures
* subdural or epidural haematomas
* parenchymal bleeds
* recent infection
* vascular anomaly
* hypertension
* current or past smoker
* high cholesterol
* family history of stroke
* migraine
* malignant/inflammatory disease
* osteoporosis
* bleeding disorde
* damaged heart valves
* pacemaker or other electrical implants
* fear of needles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline Sport Concussion Assessment Tool v5 (SCAT-5) symptom score, immediately after intervention | within 10 minutes of intervention
  Symptom numeric rating tool validated for concussion patients, 22 listed symptoms that are either present (scored 1) or absent (scored 0), minimum = 0 (good outcome), maximum = 22 (poor outcome)
Change from baseline Sport Concussion Assessment Tool v5 (SCAT-5) symptom score, 12-24 hours after intervention | 12-24 hours after intervention
  Symptom numeric rating tool validated for concussion patients, 22 listed symptoms that are either present (scored 1) or absent (scored 0), minimum = 0 (good outcome), maximum = 22 (poor outcome)
Change from baseline Sport Concussion Assessment Tool v5 (SCAT-5) symptom severity, immediately after intervention | within 10 minutes of intervention
  Symptom numeric rating tool validated for concussion patients, 22 listed symptoms that are scored from 0 (absent) to 6 (worst imaginable), minimum = 0 (good outcome), maximum = 132 (poor outcome)
Change from baseline Sport Concussion Assessment Tool v5 (SCAT-5) symptom severity, 12-24 hours after intervention | 12-24 hours after intervention
  Symptom numeric rating tool validated for concussion patients, 22 listed symptoms that are scored from 0 (absent) to 6 (worst imaginable), minimum = 0 (good outcome), maximum = 132 (poor outcome)
Change in baseline Cervical Range of Motion, immediately after intervention | within 10 minutes of intervention
  Cervical Active Range in flexion, extension, bilateral side flexion, bilateral rotation, measured in degrees using a CROM (Cervical Range of Motion) tool that measures multidirectional movement, each of the 6 ranges will be reported on their own in degrees and the 6 will also be added together for a total range measurement in degrees
Change in baseline pain score with Cervical Range of Motion, immediately after intervention | within 10 minutes of intervention
  Pain Rating Scale at end of range flexion, extension, bilateral side flexion, bilateral rotation (as measured in Outcome 5), scored 0 (no pain) - 10 (worst pain imaginable), 0 = best outcome, 10 = worst outcome, total score for all 6 movements will be computed out of 60 (0=best, 60=worst)
Change in baseline pain score with Cervical Range of Motion, 12-24 hours after intervention | 12-24 hours after intervention
  Pain Rating Scale at end of range flexion, extension, bilateral side flexion, bilateral rotation (as measured in Outcome 5), scored 0 (no pain) - 10 (worst pain imaginable), 0 = best outcome, 10 = worst outcome, total score for all 6 movements will be computed out of 60 (0=best, 60=worst)
Change in baseline of Pain Pressure Threshold (the smallest amount of pressure that evokes pain) as measured using a pressure algometer, immediately after baseline | within 10 minutes of intervention
  The pressure algometer is applied to the test muscle (in this case bilateral upper fibres trapezius, levator scapulae, suboccipital group and cervical multifidus at the base of the neck) and pressure is applied incrementally until pain is reported, the outcome is the least amount of pressure (in kilograms) applied over a muscle that evokes pain (lowest = 0 kg, higher values are better outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Margo Mountjoy, MD, Principal Investigator — Adjunct Professor
Locations (3):
- Canada (3):
  - Eramosa Physiotherapy - Elora, Elora, Ontario
  - Eramosa Physiotherapy - Bullfrog Mall, Guelph, Ontario
  - Health and Performance Centre, Guelph, Ontario

IPD SHARING:
Plan to Share IPD: No